CLINICAL TRIAL: NCT04014101
Title: A Single Arm Pilot Study of Programmed Cell Death Protein 1 Antibody (PD-1# SHR-1210 Combined With Apatinib Mesylate in Patients With Advanced-Stage Hepatocellular Carcinoma
Brief Title: SHR-1210 Plus Apatinib in Patients With Advanced-Stage Hepatocellular Carcinoma
Acronym: SHR-1210
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSGW-PD-1210
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; spartalizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210+ apatinib (Experimental): SHR-1210 was administered intravenously (without prophylaxis) at a fixed dose of 200 mg for 3 mg/kg for subjects with a baseline weight <50 kg. Each infusion for 30 min (not less than 20 min, no more than 60 min), once every 2 weeks, 1 cycle every 4 weeks, the cumulative longest medication period is 2 years; Apatinib was taken orally after meals, once a day, for continuous medication, and 1 cycle every 4 weeks.
  Interventions: Drug: SHR-1210; Drug: apatinib

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 is a humanized anti-PD-1 IgG4 monoclonal antibody
  Other Names: Anti-PD-1 Antibody
Drug: apatinib — Apatinib is a selective VEGFR2 inhibitor.

SUMMARY:
SHR-1210 is a humanized anti-PD-1 Immunoglobulin G4 (IgG4) monoclonal antibody. This is an open- label#single center #non-randomized #Single Arm Exploratory Study . This clinical study is an investigator-initiated clinical trial(IIT) .The objective of this study is to evaluate the efficacy and safety of therapy with anti-PD-1 antibody SHR-1210 and apatinib in patients with advanced stage hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1.≥18 years old, male or female 2.Advanced liver cancer (cannot be removed or metastasized) diagnosed clinically or pathologically, at least one measurable lesion without local treatment, Child-Pugh A ;Barcelona Clinic Liver Cancer(BCLC) staging is stage B or C 3.Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 4.Patient has given written informed consent. 5.Previous treatment failure with sorafenib or rivastatin (disease of disease or toxicity) or unwillingness to accept, economically unsustainable sorafenib treatment; 6.The function of important organs meets the requirements 7.Expected survival ≥12 weeks 8.Non-surgical sterilization or women of childbearing age need to use a medically-accepted contraceptive (such as an intrauterine device, contraceptive or condom) during the study period and within 3 months after the end of the study treatment period; non-surgical sterilization Female patients of childbearing age must have a negative serum or urine human chorionic gonadotropin(HCG) test within 72 hours prior to study enrollment; and must be non-lactating; for male patients with maternal age, they should be given SHR-1210 during the trial and after the last 3 effective methods of contraception within a month.

Exclusion Criteria:

- 1.The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid Hyperfunction; patients with vitiligo; complete remission of asthma in childhood, can be included without any intervention after adulthood; asthma patients who require bronchodilators for medical intervention cannot be included); 2.The patient is using immunosuppressive agents or systemic hormonal therapy to achieve immunosuppressive purposes (agents amount > 10 mg / day of prednisone or other therapeutic hormones), and continue to use within 2 weeks before enrollment; 3.Have clinical symptoms or disease that are not well controlled 4.Significant clinically significant bleeding symptoms or a clear bleeding tendency within 3 months prior to randomization 5.Arterial/venous thrombosis in the first 6 months of randomization 6.According to the investigator, the patient has other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, and serious laboratory abnormalities.，with family or social factors, it will affect the safety of patients.

7.Liver tumor burden greater than 50% of the total liver volume, or patients who have previously undergone liver transplantation;Known for a history of central nervous system metastasis or hepatic encephalopathy;Severe allergic reactions to other monoclonal antibodies;

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard

SECONDARY OUTCOMES:
Progression free survival(PFS) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
To the relief time (TOR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Duration of relief(DOR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Disease Control Rate (DCR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
9-month survival rate | 9-month
12-month survival rate | 12-month
Overall survival (OS) | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided